CLINICAL TRIAL: NCT03987230
Title: Comfort Associated With The Use Of Eyelid Cleansing Products Available For The Management Of Demodex Folliculorum
Acronym: SPANIEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40995
Record Dates: First submitted 2019-06-05; First posted 2019-06-14 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Each participant receives 6 different interventions in random order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Oust™ Demodex® Wipes™ (Active Comparator): Participant cleans eyelids with Oust™ Demodex® Wipes™
  Interventions: Other: Oust™ Demodex® Wipes™
- I-LID N LASH PLUS® Eyelid Cleanser (Active Comparator): Participant cleans eyelids with I-LID N LASH PLUS® Eyelid Cleanser
  Interventions: Other: I-LID N LASH PLUS® Eyelid Cleanser
- Blephadex Lid Wipes (Active Comparator): Participant cleans eyelids with Blephadex Lid Wipes
  Interventions: Other: Blephadex Lid Wipes
- Eye Cleanse Lid Wipes (Active Comparator): Participant cleans eyelids with Eye Cleanse Lid Wipes
  Interventions: Other: Eye Cleanse Lid Wipes
- Blephademodex (Active Comparator): Participant cleans eyelids with Blephademodex
  Interventions: Other: Blephademodex
- Sensitive Eyes® Plus Saline Solution (Placebo Comparator): Participant cleans eyelids with Sensitive Eyes® Plus Saline Solution
  Interventions: Drug: Sensitive Eyes® Plus Saline Solution

INTERVENTIONS:
Drug: Sensitive Eyes® Plus Saline Solution — Sensitive Eyes® Plus Saline Solution
  Arms: Sensitive Eyes® Plus Saline Solution
Other: Oust™ Demodex® Wipes™ — Oust™ Demodex® Wipes™
  Arms: Oust™ Demodex® Wipes™
Other: I-LID N LASH PLUS® Eyelid Cleanser — I-LID N LASH PLUS® Eyelid Cleanser
  Arms: I-LID N LASH PLUS® Eyelid Cleanser
Other: Blephadex Lid Wipes — Blephadex Lid Wipes
  Arms: Blephadex Lid Wipes
Other: Eye Cleanse Lid Wipes — Eye Cleanse Lid Wipes
  Arms: Eye Cleanse Lid Wipes
Other: Blephademodex — Blephademodex
  Arms: Blephademodex

SUMMARY:
This aim of this study to quantify the subjective ocular awareness of different eyelid cleansing wipes available for the management of Demodex folliculorum.

ELIGIBILITY:
Inclusion Criteria:

1. Is between the ages of 18 to 60 and has the full legal capacity to volunteer;
2. Has read and signed an informed consent letter;
3. Agrees to refrain from the use of ocular lubricants during the study period;
4. Agrees to not to use eye-related cosmetics for upcoming study visits
5. Is willing to use the study products
6. Is willing and able to follow instructions regarding study procedures and maintain the appointment schedule;
7. Has corneal sensitivity within physiological limits.

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Is a contact lens wearer (due to reduced corneal sensitivity);
3. Has any known active* ocular disease and/or infection; including moderate and severe dry eye (OSDI ≥ 23);
4. Has a systemic (such as diabetes, thyroid disease, rheumatoid arthritis) or ocular condition (such as glaucoma) that in the opinion of the investigator may affect a study outcome variable;
5. Is using any systemic or topical medications (such as glaucoma drops, antibiotics, anti-inflammatory) that in the opinion of the investigator may affect a study outcome variable;
6. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study (such as fluorescein dye to highlight structures of the eye and used regularly in optometric practice) and study products in this study;
7. Is pregnant, lactating or planning a pregnancy at the time of enrolment; (due to the possibility of fluctuating vision as a consequence of variation in hormone levels);8
8. Has undergone refractive error surgery (e.g. LASIK, PRK);
9. Is a smoker (as smoking reduces tear film stability) * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye (Ocular Surface Disease Index, OSDI<23/100) are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Participant's Subjective discomfort - Baseline | Baseline
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 0 seconds after application | Immediately after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 15 seconds after application | 15 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 30 seconds after application | 30 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 45 seconds after application | 45 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 60 seconds after application | 60 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 75 seconds after application | 75 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 90 seconds after application | 90 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 105 seconds after application | 105 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 120 seconds after application | 120 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 135 seconds after application | 135 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 150 seconds after application | 150 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 165 seconds after application | 165 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 180 seconds after application | 180 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 195 seconds after application | 195 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 210 seconds after application | 210 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 225 seconds after application | 225 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 240 seconds after application | 240 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 255 seconds after application | 255 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 270 seconds after application | 270 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 285 seconds after application | 285 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 300 seconds after application | 300 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 330 seconds after application | 330 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 360 seconds after application | 360 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 390 seconds after application | 390 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 420 seconds after application | 420 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 450 seconds after application | 450 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 480 seconds after application | 480 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 510 seconds after application | 510 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 540 seconds after application | 540 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 570 seconds after application | 570 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Participant's Subjective discomfort - 600 seconds after application | 600 seconds after application
  Rate the intensity of participant's ocular discomfort (0 is no discomfort, 10 is maximal discomfort)
Time to comfortably open the eyes after the application of eyelid cleansing wipe | Between 0 and 600 seconds after application
  Time to comfortably open the eyes after the application of eyelid cleansing wipe in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No